CLINICAL TRIAL: NCT07241169
Title: A Preliminary Clinical Study on the Safety and Efficacy of the Gene Replacement Drug ZVS106e in the Treatment of Hereditary Retinal Degeneration (IRDs) Caused by ABCA4 Biallelic Mutations
Brief Title: The Safety and Efficacy of ZVS106e in the Treatment of IRDs Caused by Biallelic Mutations in ABCA4
Acronym: ZVS106e
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingjiong Zhang, PI, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYA-2025-002
Record Dates: First submitted 2025-09-29; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stargardt
Keywords: ZVS106e

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All patients enrolled in the study will receive a single subretinal injection of ZVS106e in one eye
  Interventions: Drug: ZVS106e

INTERVENTIONS:
Drug: ZVS106e — ZVS106e is A colorless, clear and transparent liquid, containing two active ingredients, ZVS106E-A and ZVS106E-B. The viral vectors used for both active ingredients are rAAV8
  Other Names: rAAV8

SUMMARY:
To evaluate the preliminary safety of monocular and single subretinal injection of ZVS106e injection in the treatment of patients with hereditary retinal degeneration (ABCA4-IRDS) caused by ABCA4 biallelic mutations.

DETAILED DESCRIPTION:
The main research objective: To evaluate the preliminary safety of single subretinal injection of ZVS106e injection in one eye for patients with hereditary retinal degeneration (ABCA4-IRDS) caused by biallelic mutations in ABCA4. Secondary research objective: To preliminarily explore the clinical efficacy of ZVS106e injection in the treatment of patients with hereditary retinal degeneration (ABCA4-IRDS) caused by ABCA4 biallelic mutations. The purpose of the exploratory study is to evaluate the improvement of retinal structure and visual function in non-injection eyes compared to the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥8 years old;
2. Patients diagnosed with hereditary retinal degeneration caused by ABCA4 biallelic mutations through genetic testing, and without other ophthalmic genetic diseases;
3. The target eye must meet the following requirements: the best corrected visual acuity is 0.5 to 2.0 LogMAR (including 0.5 and 2.0 LogMAR, equivalent to the decimal visual acuity index up to 0.3);
4. The subject and his or her spouse agree to take effective contraceptive measures during the trial period and for at least one year after administration.
5. Voluntarily participate in clinical trials and sign informed consent forms, and be able to complete all trial processes as required by the protocol.

Exclusion Criteria:

1. The researchers determined that the target eye currently has or has previously had other macular lesions such as retinal schisis or epiretinal membrane. Or have other eye diseases that may hinder the surgery or interfere with the interpretation of the study endpoint;
2. Having received drug treatment that may affect the observation of the trial within the three months prior to screening;
3. The target eye has undergone the following intraocular surgeries: retinal repositioning and vitrectomy;
4. There are known eye/visual diseases, disorders or lesions that cause or are related to vision loss, or whose related treatments or therapies are known to cause or are related to vision loss;
5. Having suffered from a viral infectious disease that may affect the efficacy and safety evaluation of the investigational drug or having received an antiviral vaccine within one month prior to enrollment;
6. Systemic medications that are currently in use or may be required to cause eye toxicity, such as psoralen, risselinic acid or tamoxifen, etc.
7. Known to be allergic to the drugs planned to be used in the study;
8. Suffering from poorly drug-controlled hypertension: systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg;
9. The following laboratory test abnormalities have clinical significance:

   Liver function: Chronic liver disease, elevation of ALT or AST >2 times the upper limit of the normal value; Those with abnormal coagulation function (prothrombin time ≥ 3 seconds above the upper limit of the normal value, activated partial thromboplastin time ≥ 10 seconds above the upper limit of the normal value); Serum virological examination: Positive for active hepatitis B, hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or syphilis antibody;
10. There is any past or current medical history that may affect the safety of the trial or the in vivo process of the drug, especially a history of diseases such as cardiovascular, liver, kidney, endocrine, digestive tract, lung, nervous, hematological, tumor, immune or metabolic disorders that the investigators consider to have clinical significance;
11. Those who have participated in any clinical trials of drugs or medical devices within the three months prior to screening;
12. Pregnant or lactating women; According to the researcher's judgment, those who are deemed unsuitable to participate in this clinical trial for other reasons

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of subretinal injection of ZVS106e solution | 52 weeks post-treatment
  Types, severity, and incidence of adverse events (AE) and serious adverse events (SAE) in the eyes and throughout the body within 52 weeks post-treatment, including dose-limiting toxicities (DLT) during the dose escalation phase.

SECONDARY OUTCOMES:
Change from baseline in best-corrected visual acuity (BCVA) | 52 weeks post-treatment
  Change in best-corrected visual acuity (BCVA) of the treated eye at 52 weeks compared to baseline.
Change from Baseline in Visual function metrics | 52 weeks post-treatment
  Treatment outcomes for visual function metrics include changes from baseline in LLVA, dynamic visual field, microperimetry, FST, contrast sensitivity, color vision, and mfERG; as well as changes from baseline in the NEI-VFQ-25 score reported by the participants.
Change from Baseline in OCT | 52 weeks post-treatment
  Compare changes in retinal morphology and alterations in cell layers of the retina before and after drug administration.
Change from Baseline in multi-luminance mobility test (MLMT) | 52 weeks post-treatment
  MLMT was assessed using both eyes at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night).
Change from Baseline in Fundus autofluorescence (FAF) | 52 weeks post-treatment
  Compare the atrophy of the RPE/ photoreceptor complex in the subjects before and after administration

OTHER OUTCOMES:
Change from Baseline in Michigan Retinal Degeneration Questionnaire (MRDQ) | 52 weeks post-treatment
  Compare the improvement effects of vision-related anxiety in patients before and after administration
Change from Baseline in multiluminance shape discrimination test (MLSDT) score | 52 weeks post-treatment
  The improvement of the recognition ability for objects of different sizes under different brightness conditions before and after administration was compared. The higher the score, the stronger the shape recognition ability

CONTACTS AND LOCATIONS:
Overall Officials: qingjiong zhang, M.D, Study Director — PI; lin Lv, M.D, Principal Investigator — PI

IPD SHARING:
Plan to Share IPD: No